CLINICAL TRIAL: NCT02029963
Title: The Efficacy of Repetitive Transcranial Magnetic Stimulation in Relapse Prevention of Major Depressive Disorder
Brief Title: Can Magnetic Brain Stimulation Help Prevent Relapse in Depression?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful in obtaining recruitment
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2013:178
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cluster rTMS (Experimental): Two weeks of daily repetitive Transcranial Magnetic Stimulation (total of 10 rTMS sessions), six months following completion of regular six-week rTMS treatment.
  Interventions: Device: Transcranial Magnetic Stimulation (rTMS)
- Taper rTMS (Experimental): Immediately following completion of regular six-week repetitive Transcranial Magnetic Stimulation treatment, patients in this group will receive three sessions of rTMS a week for two weeks followed by two sessions of rTMS a week for two weeks (total of 10 rTMS sessions tapered in 4 weeks)
  Interventions: Device: Transcranial Magnetic Stimulation (rTMS)
- Treatment as Usual (Experimental): Following their last session of regular six-week rTMS treatment, patients in this group will follow an individually-tailored maintenance plan as determined by their own psychiatrist or primary care provider
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (rTMS) — A non-invasive method for brain stimulation
  Arms: Cluster rTMS; Taper rTMS
Behavioral: Treatment as Usual — An individually-tailored maintenance plan as determined by a psychiatrist or primary care provider
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to investigate the use of repetitive transcranial magnetic stimulation (rTMS) in helping to prevent relapse in major depressive disorder. rTMS is known to be an effective treatment for major depressive disorder, but there is also evidence that it may be effective in the maintenance of remission following treatment. However, it is not yet clear what maintenance strategy will yield the best outcome in preventing relapse.

In this study, eligible patients who have finished one full course of rTMS for treatment of major depression will be randomized into three groups: (i) cluster rTMS, (ii) taper rTMS, and (iii) treatment as usual. The 'cluster rTMS' group will receive two weeks to daily rTMS six months after the completion of their regular rTMS treatment, the 'taper rTMS' group will receive three sessions a week for two weeks followed by two sessions a week for two weeks immediately following their regular rTMS treatment, while the 'treatment as usual' group will receive standard follow-up care from their own psychiatrist and/or primary care doctor.

The investigators hypothesize that the group with cluster treatment will show significantly lower relapse rates in depressive symptoms as compared to the other groups.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy of rTMS to the dorsolateral prefrontal cortex (dlPFC) as a maintenance therapy following standard rTMS treatment in major depressive disorder.

A total of 45 patients will be recruited for this study. Patients who have completed a standard six-week rTMS treatment for major depressive disorder will be randomly assigned to one of the three groups: cluster rTMS, taper rTMS, and treatment as usual. Patients in the 'cluster' group will receive two weeks of daily rTMS (10 rTMS sessions) six months after completing their rTMS treatment. Patients in the 'taper' group will receive rTMS immediately after completing rTMS treatment and the frequency of the sessions will be tapered as follows: three sessions a week for two weeks, and then two sessions a week for two weeks. The maintenance plan for patients in 'treatment as usual' group will be decided individually and may include any or all of the following: continue or start on medication, start psychotherapy and/or follow-up visits with psychiatrist or primary care provider.

Each session of rTMS will be identical: lasting about one hour and consisting of 3000 high frequency (10 Hz) pulses. After finishing their last session of rTMS treatment, all patients will be seen by the rTMS psychiatrists bi-monthly for one year. Each visit will last approximately half an hour during which time the Hamilton Depression (Ham-D) Scale will be administered.

Given the high relapse rates following rTMS treatment for depression, the investigators hope that results from this study will be very helpful to patients suffering from major depressive disorder in improving their quality of life by reducing their rate of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Major Depressive Disorder
* Patients who are not actively receiving any psychotherapy
* Patients who are on no or only one antidepressant

Exclusion Criteria:

* History of a psychotic episode
* History of neurological illness
* Previous head injury
* Active alcohol or substance abuse
* History of seizure disorders
* Currently pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptom severity | One year with bi-monthly measurements
  Changes in depressive symptoms will be measured through administration of the Hamilton Depression (Ham-D) Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Modirrousta, MD PhD, Principal Investigator — Saint Boniface General Hospital
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada